CLINICAL TRIAL: NCT03676062
Title: Kronik Bel Ağrılı Bireylerde Yoga ve Spinal Stabilizasyon Egzersizlerinin Ağrı, Fonksiyon ve Stres Üzerine Etkisinin Karşılaştırılması
Brief Title: The Effect of Yoga and Stabilization Exercise in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Muzeyyen Oz, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GO15/81
Record Dates: First submitted 2018-08-06; First posted 2018-09-18 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Chronic Low Back Pain
Keywords: exercise, pain, yoga
MeSH Terms: conditions — Motor Activity; Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- stabilization exercise group (Active Comparator): Spinal stabilization exercise were applied all patients additional with hotpack, TENS application in this group accompanied by physiotherapist.
  Interventions: Other: exercise
- yoga group (Active Comparator): Yoga program were applied all patients in this group accompanied by physiotherapist. Sessions included selected breathing exercises, warm up, asana and relaxation.
  Interventions: Other: exercise
- home exercise group (Active Comparator): Home exercise were applied all patients in this group supervised, controlled by physiotherapist every week.To make compliance easier for patients; a booklet including suggestions to prevent low back pain and description of exercises, were given. Prescribed exercises were selected in this booklet and checked&progressed in each control sessions.
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — All exercises programs applied three sessions per week, totally six week.

SUMMARY:
Identification of the effects of yoga, stabilization exercise and home exercise approaches on pain, function,stress and quality of life in individuals with low back pain.

DETAILED DESCRIPTION:
44 patients participating in the study were divided three groups. The patients in the stabilization exercise group were instructed to perform hotpack, Trans-cutaneous Electric Nerve Stimulation (TENS) and spinal stabilization exercises, the patients in the yoga group were instructed to perform yoga program consisting of breathing, relaxation and flexibility exercises. The patients in the home exercise group were instructed to perform stabilization exercise. The severity of the pain evaluated through visual analog scale, functional status and quality of life evaluated through Oswestry Disability Index(ODI), Nottingham Health Profile (NHP), respectively. Assessments were repeated before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must be pain at least 3 months
* Must be visual analog scale rating 3 or more

Exclusion Criteria:

* History of any lumbar spine surgery
* Severe/progressive scoliosis
* Spinal stenosis
* Spondylolisthesis
* Cancer
* Diabetes
* Metabolic syndrome
* History of exercise programs or yoga at least 12 weeks before the onset of study

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Changes in pain severity | change from baseline in pain severity at 6 weeks.
  Patients' average resting and activity pain intensities assessed by Visual Analog Scale.
  The visual analog scale is an 11-point scale ranging from 0 to 10, in which 0 defines absence of pain and 10 describes unbearable pain. Participants asked to rate the average pain levels a horizontal 10 cm straight line on a white sheet from, before and after treatment.

SECONDARY OUTCOMES:
Changes in quality of life | Change from baseline in life quality levels at 6 weeks.
  Health-related quality of life assessed by Nottingham Health Profile (NHP). The NSP contain 38 questions in 6 subareas: pain, physical abilities, energy level, sleep, social isolation and emotional reaction. The scores range from 0 to 100, with each question assigned a weighted value; the sum of all weighted values in a given subarea adds up to 100. Lower scores denoting a better quality of life.
Changes of functional status | change from baseline in functional status at 6 weeks
  Patient's permanent functional disability measured by Oswestry Disability Index. The scale is considered the 'gold standard' of low back functional outcome tools. This scale contain questions related to functional activities of pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life, social life and travelling.Interpretation of scale are 0% to 20% for minimal disability, 21% to 40% for moderate disability, 41 % to 60 % for severe disability 61% to 80 % for crippled and 81 % to 100 % Bed-bound.
Changes of stress level | change from baseline in stress level at 6 weeks
  Patients' stress levels were measured with State Trait Anxiety Inventory. State anxiety scale questions how does a person feel in a given moment and situation, mean while trait anxiety scale questions how does a person usually feel without depending on situation and moment. Scale contain 40 questions, minimum and maximum score 20-80, respectively. Scores below 36 accepted as "no-anxiety", between 37-42 accepted as "low-anxiety", 42 and above accepted as "high-anxiety.
Changes of stress related biomarkers | change from baseline in serum level at 6 weeks
  Venous blood samples were taken from antecubital area between 08.30-09.00 am and stress related markers (DHEA(S) and cortisol) were analyzed. All analyses were performed in the same laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Müzeyyen ÖZ, MSc, Principal Investigator — Hacettepe University; Özlem ÜLGER, Asc. Proff, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Health Sciences Faculty, Ankara, Altındag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Inani SB, Selkar SP. Effect of core stabilization exercises versus conventional exercises on pain and functional status in patients with non-specific low back pain: a randomized clinical trial. J Back Musculoskelet Rehabil. 2013;26(1):37-43. doi: 10.3233/BMR-2012-0348. PMID 23411647
- [Result] Nambi GS, Inbasekaran D, Khuman R, Devi S, Shanmugananth, Jagannathan K. Changes in pain intensity and health related quality of life with Iyengar yoga in nonspecific chronic low back pain: A randomized controlled study. Int J Yoga. 2014 Jan;7(1):48-53. doi: 10.4103/0973-6131.123481. PMID 25035607
- [Result] Shirado O, Doi T, Akai M, Hoshino Y, Fujino K, Hayashi K, Marui E, Iwaya T; Japan Low back-pain Exercise Therapy Study; Investigators Japanese Orthopaedic Association; Japanese Society for Musculoskeletal Rehabilitation; Japanese Clinical Orthopaedic Association. Multicenter randomized controlled trial to evaluate the effect of home-based exercise on patients with chronic low back pain: the Japan low back pain exercise therapy study. Spine (Phila Pa 1976). 2010 Aug 1;35(17):E811-9. doi: 10.1097/BRS.0b013e3181d7a4d2. PMID 20628332
- [Result] Cho I, Jeon C, Lee S, Lee D, Hwangbo G. Effects of lumbar stabilization exercise on functional disability and lumbar lordosis angle in patients with chronic low back pain. J Phys Ther Sci. 2015 Jun;27(6):1983-5. doi: 10.1589/jpts.27.1983. Epub 2015 Jun 30. PMID 26180363